CLINICAL TRIAL: NCT07276659
Title: The Contribution of Scenario Writing to Learning Stoma Care in Nursing Education: A Mixed-Methods Quasi-Experimental Intervention Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: hatice akaltun (Other)
Responsible Party: Sponsor-Investigator, hatice akaltun, Lecturer (PhD) in Nursing, Yuzuncu Yil University
Organization: Yuzuncu Yil University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: VYYU-SBF-HAKALTUN-002
Record Dates: First submitted 2025-11-29; First posted 2025-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Stoma Care Education in Nursing Students
Keywords: Stoma Care; Scenario-Based Learning; Nursing Education

STUDY DESIGN:
Intervention Model Description: Two-arm quasi-experimental design with an intervention group receiving scenario-writing-based stoma care education and a passive control group
Masking Description: No masking was applied; participants and investigators were aware of group assignments
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Scenario-Based Stoma Care Education (Experimental): Participants in the intervention arm will receive an 8-week scenario-based stoma care education program.
  The intervention includes:
  * 4 weeks of scenario writing sessions,
  * 4 weeks of role-play/dramatization in the skills laboratory,
  * Structured feedback by the instructor. No additional theoretical lecture will be provided. Participants complete pre-test and post-test assessments, and qualitative focus group interviews will be conducted after completion of the intervention.
  Interventions: Behavioral: Scenario-Based Stoma Care Education
- Control Group (No Intervention): Participants in the control arm will not receive any additional education or training.
  They will complete the same pre-test and post-test assessments as the intervention group.
  No scenario writing or role-play activities will be administered.

INTERVENTIONS:
Behavioral: Scenario-Based Stoma Care Education — A structured scenario-writing and role-play-based educational program delivered over 8 weeks. Students develop stoma care scenarios, present them, and perform role-play using simulated patients and a skills laboratory environment. The intervention includes scenario writing sessions (4 weeks) and stoma care role-play practice using manikins and real materials (4 weeks), followed by structured educator feedback.
  Arms: Scenario-Based Stoma Care Education

SUMMARY:
This study aims to evaluate the effectiveness of scenario writing and role-play-based learning on nursing students' knowledge related to stoma care. The study uses a mixed-methods, quasi-experimental design including an intervention and a control group. Students in the intervention group participate in an eight-week scenario-based learning program consisting of scenario writing, dramatization (role-play), and structured feedback sessions. The control group receives no additional educational activity beyond the standard curriculum. Stoma care knowledge is assessed using a pre-test administered on October 27, 2025, and a post-test administered on December 22, 2025. In addition, qualitative data are collected from intervention-group participants through semi-structured focus group interviews to explore changes in confidence, perceived skills, and learning experiences. The goal of the study is to determine whether scenario-based learning strengthens the acquisition of stoma care knowledge and enhances students' educational experiences.

DETAILED DESCRIPTION:
This mixed-methods quasi-experimental study investigates the impact of scenario-based learning on nursing students' acquisition of stoma care knowledge. Third-year nursing students who previously completed the surgical nursing course were eligible for participation. The intervention group engaged in an eight-week Scenario-Based Stoma Care Learning Program, which included (1) preparation and writing of clinical scenarios, (2) dramatization and role-play activities using simulated clinical environments, and (3) structured instructor-guided feedback. The control group did not receive any additional training and completed only the pre-test and post-test assessments.

The pre-test measuring stoma care knowledge was administered on October 27, 2025. The post-test was administered on December 22, 2025, following completion of all scenario-based learning sessions. After the educational intervention, qualitative data were collected from the intervention group through focus group interviews using a COREQ-aligned semi-structured interview guide. Qualitative data aim to explore changes in participants' confidence, perceived skills, learning processes, and their experience with scenario writing and role-play.

The study's primary objective is to determine whether scenario-based learning improves students' stoma care knowledge. Secondary objectives include understanding how scenario writing and dramatization influence students' confidence, engagement, and perceived competence in performing stoma care.

ELIGIBILITY:
Inclusion Criteria:

* Being a 3rd-year undergraduate nursing student in the Nursing Department.
* Having successfully completed the Surgical Nursing course in the 2nd year.
* Voluntarily agreeing to participate in the study and providing informed consent.

Exclusion Criteria:

* Students who did not pass the Surgical Nursing course.
* Students who have previously received professional stoma care training.
* Students who complete the data collection forms incompletely.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-10-27 (Actual); Primary Completion 2025-12-22 (Estimated); Study Completion 2025-12-22 (Estimated)

PRIMARY OUTCOMES:
Stoma Care Knowledge Score | Baseline (Week 0) and Post-intervention (Week 8)
  Change in students' stoma care knowledge score from pre-test to post-test. Knowledge will be measured using a 20-item Stoma Care Knowledge Questionnaire developed by the research team. Scores range from 0 to 20, with higher scores indicating greater knowledge. The primary analysis will compare post-test scores between the intervention and control groups, adjusting for baseline knowledge.

SECONDARY OUTCOMES:
Qualitative Themes Related to Students' Perceived Confidence and Skill Development | Immediately after completion of the 8-week intervention (same week as the post-test).
  Semi-structured focus group interviews will be conducted with participants in the intervention group after completion of the 8-week program. Qualitative analysis (thematic analysis) will explore changes in perceived confidence, perceived competence, motivation for practice, and learning experiences related to scenario writing and role-play activities. Themes will be identified using coded transcripts analyzed with MAXQDA by two independent researchers.

CONTACTS AND LOCATIONS:
Overall Officials: hatice akaltun, PhD, Principal Investigator — Yuzuncu Yil University
Locations (1):
- Van Yuzuncu Yil Univeristy, Van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared because the ethical approval does not permit disclosure of identifiable or de-identified participant-level data